CLINICAL TRIAL: NCT06171893
Title: The Multicentre Wavy Stress Study: Assessing the Effect of the 'Wavy' Application, on Stress and Burden of Disease in Women With INOCA Caused by Vasospasms.
Brief Title: Assessing the Effect of the 'Wavy' Application, on Stress and Burden of Disease in Women With INOCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: VieCuri Medical Centre (Other); The Elisabeth-TweeSteden Hospital (Other); Maastricht University Medical Center (Other); Maasstad Hospital (Other); Catharina Ziekenhuis Eindhoven (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Health Holland (Other); Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: .NL77493.091.21
Record Dates: First submitted 2023-11-28; First posted 2023-12-15 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Stress; Ischemia; Vasospasm, Coronary; Vasomotor; Spasm; Angina, Stable; Prinzmetal Angina
MeSH Terms: conditions — Ischemia; Coronary Vasospasm; Spasm; Angina, Stable; Angina Pectoris, Variant

STUDY DESIGN:
Intervention Model Description: A single-arm, controlled, multicentre trial, will be conducted to validate to study objective. The study is divided into five iterative substudies of which the first four are aimed towards improving the application, based on the quantitative data from the smartwatch and the qualitative feedback of the users whilst also validating the recent version through assessing the interim study outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control vs intervention (Experimental): Each subject will take part in a four-week control period, followed by a four-week intervention period.
  Interventions: Behavioral: Wavy stress application

INTERVENTIONS:
Behavioral: Wavy stress application — The intervention consists of the application named Wavy. Wavy uses artificial intelligence and the user's feedback to detect stress increasingly more efficient over time. This provides not only real-time feedback on an individual's stress level but also helps the patient to calm down using music guided relaxation. It does so with a music filter, allowing the participant to listen to music where the stress level determines the quality of the music.
  Thus, relaxing is rewarded by improving the experience. In this process, implicit learning is used to establish a habit of getting better at recognising increased stress levels and getting familiar with reducing stress levels more and more effectively.

SUMMARY:
For women that experience angina symptoms with underlying vascular spasm as the cause, stress has an aggravating role. Coping with stress is therefore included as an important pillar in dealing with this chronic disease, see the European Association of Percutaneous Cardiovascular Interventions (EACPI) consensus document on INOCA. In practice, stress management focuses on informing and identifying the role stress plays in their lives. A potential stress management tool: "Wavy" aims to help users manage stress more consciously through biofeedback. This research focuses on the effectiveness of stress management applications. The hypothesis is that the app will help to avoid the trigger stress as much as possible and thus reduce the burden of disease.

DETAILED DESCRIPTION:
Rationale: The majority of women with angina and non-obstructive coronary arteries (INOCA) do have underlying epicardial or microvascular coronary vasospasms as revealed by invasive vasomotor testing. It is well known that stress is one of the important triggers of coronary vasospasms, therefore, stress reduction is of importance to this population. 'Wavy' is a smartphone application that estimates stress levels through a collection of physiological data by smartwatches and offers music guided relaxation through bio-feedback when these levels appear too high. It is hypothesized that the use of 'Wavy' will result in less stress and consequently fewer complaints of angina pectoris.

Objective: This study sets out to assess whether incorporating Wavy in daily life results in a better quality of life as measured through the primary outcome: visual analogue scale on pain (VAS) score and secondary outcomes: perceived stress score (PSS-10) quality of life (SF-36), heart rate variability (HRV) based stress levels, and angina frequency.

Study design: Patients will be enrolled in a single-arm placebo-controlled multicentre trial, consisting of 4 weeks placebo followed by 4 weeks intervention.

Study population: The study population will consist out of 250 women from 5 cardiology centres, aged between 18 and 70, who are diagnosed with INOCA with coronary vasomotor disorders.

Intervention: The smartphone application ''Wavy'' offers music guided relaxation when stress levels, as measured by biological parameters through the wearable, are too high.

Main study parameters/endpoints: The primary study parameter is the difference between the VAS scores before and after the intervention period.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: To ensure a low burden for the participants, the trial will be executed digitally, meaning that, aside from delivering the wearables, all contact will be through online and phone contact. Over the course of approximately two months, the participant will be asked to watch an introduction video series, explaining the proper usage of Wavy Assistant, also they will be asked to wear a smartwatch, and to use a music guided relaxation for approximately 10 minutes at a time. In addition, the participants will be asked to fill out three questionnaires twice, taking approximately ninety minutes in total. Overall, the risk of the intervention is negligible. The potential benefit of the intervention is a reduction of symptoms of angina in patients through music guided relaxation, which is a natural, non-medical therapy without risk of side effects.

ELIGIBILITY:
Female participants are recruited from the cardiology outpatient clinics at the department of cardiology Radboudumc, Maastricht UMC, Catharina Hospital Eindhoven, St. Elisabeth Hospital Tilburg, Maasstad Hospital and in VieCuri MC, Venlo. All participants have must meet

Inclusion criteria:

1. Female.
2. Aged 18-70 (upper-limit, because of increased comorbidities and potential difficulties with using the technology).
3. Suffering from chronic angina pectoris.
4. Diagnosed with INOCA, documented within 2 years, with a coronary angiogram and an abnormal coronary function test (CFT), indicative of either epicardial or microvascular vasospasms.
5. Daily usage of a smartphone with an operating system equal to or higher than Android 5.0 (Lollipop) or IOS 10.0.
6. Signed written informed consent.

Excluded criteria:

1. She is not available for the assigned research period of approximately 10 weeks from May 2021 till October 2022. The application can be used during the planned holidays.
2. She is unable to participate in the stress-reducing exercise, e.g., due to hearing problems.
3. A language barrier is present.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
seattle angina questionnaire | 10 weeks
  A valid, reproducible, responsive instrument for assessing disease-specific health status among patients with coronary artery disease

SECONDARY OUTCOMES:
VAS score on pain | 10 weeks
  Visual scale of 1-100 on pain
Heart rate variability | 10 weeks
  Semi semi-continuous 30 second heart rate variabillity (hrv) derived from photoplethysmogram (PPG) signal measurements each 15 minutes
Perceived stress score | 10 weeks
  PSS-10 questionnaire, validated questionnaire indicating perceived stress
SF-36 | 10 weeks
  Quality of life questionnaire
Symptom diary | 10 weeks
  Descriptions and time labeling of experienced symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Suzette Elias-Smale, dr., Principal Investigator — Radboud University Medical Center
Locations (6):
- Netherlands (6):
  - Radboud universty medical center, Nijmegen, Gelderland
  - Maastricht UMC, Maastricht, Limburg
  - VieCuri, Venlo, Limburg
  - Catharina Hospital, Eindhoven, North Brabant
  - Elisabeth-TweeSteden Hospital, Tilburg, North Brabant
  - Maasstad Hospital, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: No